CLINICAL TRIAL: NCT00987987
Title: Amplifying Graft-versus-tumor Effect by Donor Regulatory T-cell Depletion Before Donor Lymphocytes Infusion: a Phase I/II Clinical Study
Brief Title: Amplifying Graft-Versus-Tumor Effect by Donor Regulatory T-Cell Depletion Before Donor Lymphocytes Infusion
Acronym: ILD-Treg
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Université Paris XII (Unknown); Pierre and Marie Curie University (Other)
Responsible Party: Valérie Millul, Department Clinical Research of Developpement
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P040441
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2009-09

CONDITIONS: Hematologic Neoplasms; Relapse
Keywords: hematological malignancy; allogeneic hematopoietic stem cell transplantation; donor lymphocyte infusion; antitumor immunotherapy; graft-versus-tumor effect; regulatory T cells; adult
MeSH Terms: conditions — Hematologic Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 1
  Interventions: Procedure: donor lymphocyte infusion

INTERVENTIONS:
Procedure: donor lymphocyte infusion — regulatory T cells depletion
  Other Names: regulatory T cells depletion

SUMMARY:
The investigators have previously shown that depletion of CD4+CD25+FoxP3+ regulatory T cells (Treg) enhances the alloreactivity of T lymphocytes, as attested by an accelerated GVHD after allogeneic hematopoietic stem cell transplantation (HSCT) in mice. The investigators thus propose a clinical trial to test whether Treg-depleted donor lymphocytes infusion (dDLI) could induce an improved graft-versus-tumor (GVT) effect in patients refractory to standard DLI (stdDLI) for treatment of relapse after HSCT.

DETAILED DESCRIPTION:
We have previously shown that depletion of CD4+CD25+FoxP3+ regulatory T cells (Treg) enhances the alloreactivity of T lymphocytes, as attested by an accelerated GVHD after allogeneic hematopoietic stem cell transplantation (HSCT) in mice. We thus propose a clinical trial to test whether Treg-depleted donor lymphocytes infusion (dDLI) could induce an improved graft-versus-tumor (GVT) effect in patients refractory to standard DLI (stdDLI) for treatment of relapse after HSCT.

dDLI is administered after failure of 1 or several previous stdDLI of at least 107 CD3+ cells/kg, defined after a minimal follow-up of 2 months after the last injection. The absence of previous clinical manifestations of GVHD is required to be included. To prepare dDLI, CD25+ Treg are depleted from donor leukaphereses using anti-CD25 magnetic microbeads and a CliniMACS device (MYLTENYI). In order to evidence the potential effect of dDLI, the dDLI cell dose is adjusted to be below or equal to the maximal cell dose previously received in stdDLI. No comparison is planned in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Hematological malignancy except chronic myeloid leukaemia.
* Previous allogeneic hematopoietic stem cell transplantation.
* Relapse diagnosed at the molecular, cytogenetic, or cytological level.
* Failure of a previous stdILD or inclusion in first intention if progressive disease.
* Age > 18 years and < 70 years at the time of inclusion.
* Performance status considered on the score ECOG < 2.
* Life expectation 1-month-old superior.
* Signed written informed consent.
* Negative HCG in the 7 days preceding the inclusion for women in age of procreation.
* Membership of the French national insurance.

Exclusion Criteria:

* Chronic myeloid leukemia
* Grade >II acute GVHD or chronic extensive GVHD at the time of inclusion.
* Patient receiving an immunosuppressive treatment for GVHD treatment at the time of inclusion.
* Dysfunction of liver (ALAT/ASAT > 5 N, or bilirubin > 50 µM), or of the renal function (creatinine clearance < 30 ml / min).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2005-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Incidence of "severe" GHVD (grade >II) following dDLI should be inferior to 40%. | 4 weeks after dDLI

SECONDARY OUTCOMES:
The incidence of GVHD of any grade after dDLI | during the 12 months
The anti-tumoral efficiency of dDLI to treat the relapse of the hematological malignancy | during the 12 months
The survival and the survival without disease after dDLI | during the 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Maury, MD Ph, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Henri Mondor, Créteil, France

REFERENCES:
- [Result] Maury S, Lemoine FM, Hicheri Y, Rosenzwajg M, Badoual C, Cherai M, Beaumont JL, Azar N, Dhedin N, Sirvent A, Buzyn A, Rubio MT, Vigouroux S, Montagne O, Bories D, Roudot-Thoraval F, Vernant JP, Cordonnier C, Klatzmann D, Cohen JL. CD4+CD25+ regulatory T cell depletion improves the graft-versus-tumor effect of donor lymphocytes after allogeneic hematopoietic stem cell transplantation. Sci Transl Med. 2010 Jul 21;2(41):41ra52. doi: 10.1126/scitranslmed.3001302. PMID 20650872